CLINICAL TRIAL: NCT02167646
Title: Bilaterally Innervated Sensory Dorsal Digital Flaps for Sensory Reconstruction of the Fingers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSChen10512; HBTS14-01502 (Other: Ethics Committee of Hebei)
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2012-02

CONDITIONS: Soft Tissue Injuries
Keywords: Soft tissue defect; dorsal branch of the digital nerve; dorsal branch of the digital artery; dorsal digital flap
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bilaterally innervated flap (Other): Two nerve branches attached with the flap for sensory reconstruction.
  Interventions: Procedure: Flap including bilateral nerve branches

INTERVENTIONS:
Procedure: Flap including bilateral nerve branches — Two nerve branches are attached with the flap for sensory coverage

SUMMARY:
Sensory coverage in the finger continues to be a challenging problem. This study reports sensory reconstruction of the fingers with the bilaterally innervated dorsal digital flaps and compares the results between the dual- and single-innervated flaps.The main evaluated outcomes are static 2-point discrimination and Semmes-Weinstein monofilament scores of the flap, fingertip pain and joint motion.

DETAILED DESCRIPTION:
Pain was given subjectively by the patient using the visual analogue scale (VAS). The VAS consists of a 10 cm line that was grouped into mild (0-3 cm), moderate (4-6 cm) and severe (7-10 cm). Tinel's sign was rated as the following: grade 1=none; grade 2=mild, slight tingle; grade 3=moderate, very uncomfortable; and grade 4=severe, patient unable to use hand because of any stimulation of the neuroma.

ELIGIBILITY:
Inclusion Criteria:

* a soft-tissue defect in the areas where sensory return was considered important ●a defect with exposed bone or tendon in one finger
* the defect associated with the transected digital nerves in both sides
* a defect greater than 1.5 cm
* a patient aged 15 to 60 years

Exclusion Criteria:

* injuries to the dorsum of the finger or to the course of the vascular pedicle that precluded its use as the donor
* injuries to the dorsal branches of the digital nerves that precluded its use as donor nerves attached with the flap
* a defect less than or equal to 1.5 cm
* patient age < 15 years or > 60 years

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Static 2PD test | 18 months to 24 months after surgery
  We use a Disk-Criminator to test two nearby points when touching the flap

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Chen C, Tang P, Zhang X. The dorsal homodigital island flap based on the dorsal branch of the digital artery: a review of 166 cases. Plast Reconstr Surg. 2014 Apr;133(4):519e-529e. doi: 10.1097/PRS.0000000000000016. PMID 24675204
- [Derived] Chen C, Tang P, Zhao G. Bilaterally innervated dorsal digital flap for sensory reconstruction of digits. Injury. 2014 Dec;45(12):2018-24. doi: 10.1016/j.injury.2014.09.012. Epub 2014 Sep 22. PMID 25304161